CLINICAL TRIAL: NCT04090827
Title: A Mixed Methods RCT Evaluating a Telehealth-based Nurse-led Transition Intervention in Combination With Access to a CHD Website, vs. the CHD Website Alone, on Preparing Rural-based Adolescents Living With CHD to Successfully Transition From Pediatric to Adult Cardiology Care
Brief Title: The Transitioning Rural Adolescents to Adult Care Study
Acronym: TRAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00074194
Record Dates: First submitted 2019-06-26; First posted 2019-09-16 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Transition; Congenital Heart Defect
Keywords: transition; Congenital heart disease; education; adolescence
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Nurse-led transition intervention and access to the iHeartChange website
  Interventions: Other: Nurse-led transition intervention and access to the iHeartChange website

INTERVENTIONS:
Other: Nurse-led transition intervention and access to the iHeartChange website — Elements of the transition interventions include: (i) introduction to transition and its importance, (ii) creation of a MyHealth Passport, (iii) review diagram of participant's cardiac anatomy, (iv) discussion of 3 potential future cardiac complications (v) iHeartChange website (vi) discussion of the concept of "self-management" (vii) discussion and promotion of communication skills by the adolescent with their healthcare team via the GLADD technique (Give, Listen, Ask, Decide, Do) (viii) a "3-sentence summary" about their CHD (ix) ongoing text/email support from RN

SUMMARY:
Approximately 1 in 10 teenagers lives with a chronic health condition that will require ongoing care as they enter adulthood. Birth defects of the heart, also known as congenital heart disease (CHD) are more common than any other type of birth defect and affect about 1 in 100 children, with most surviving to adulthood. However, most teenagers with CHD have little knowledge about their heart and lack confidence in talking with doctors and nurses about their health. These are essential skills when entering the adult-oriented health care system after graduating from pediatric care.

In the current study proposal our team plans to evaluate the effectiveness of delivering 1-on-1 teaching sessions for adolescents who live in smaller communities and can't easily come to Edmonton for appointments in the heart clinic. Fortunately in Alberta we have a widely available system called Telehealth that allows nurses and teens to meet by private, secure teleconferencing while hundreds of miles away. Telehealth is provided by health clinics around the province. We propose to use Telehealth in adolescents' home communities to provide these teaching sessions for 16-19 year olds with CHD who are soon going to be graduating from pediatric to adult care.

Participants who receive a nurse-led teaching session will be compared with a similar number of adolescents who are not offered a teaching session, using a questionnaire that addresses skills related to taking care of their health condition. This questionnaire will be completed on-line (or if preferred by the participant, by letter mail) 1 month and 6 month after entering the study.

Deciding which adolescents receive a nurse-led teaching session will be random, i.e. like the flip of a coin. Regardless, all participants will receive access to a website for young people with CHD called iHeartChange.

DETAILED DESCRIPTION:
PURPOSE:

The Transitioning Rural Adolescents to Adult Care (TRAAC) Study is a prospective cohort study evaluating the impact of a Telehealth-based nurse-led transition intervention in combination with access to a CHD website on preparing rural-based adolescents living with congenital heart disease (CHD) to successfully transition from pediatric to adult cardiology care.

OBJECTIVES:

The primary objective is to determine the impact of a nurse-led transition intervention in combination with access to the iHeartChange website on adolescents' knowledge of their heart [Hypothesis: the nurse-led intervention will result in superior CHD knowledge compared to baseline].

The secondary objectives are to:

(i) evaluate the impact of the nurse-led intervention on adolescents' self-efficacy [Hypothesis: the nurse-led intervention will result in superior self-efficacy compared to baseline],

(ii) evaluate the impact of the nurse-led intervention on adolescents' self-management skills [Hypothesis: the nurse-led intervention will result in superior self-management skills compared to baseline].

(iii) measure frequency of iHeartChange use by participants

RESEARCH METHOD:

Participants will be recruited through the Stollery Children's Hospital Outreach Pediatric Cardiology clinics. After discussion with the Research Coordinator, the participant will be emailed an online consent form, and baseline questionnaires through REDCap as well as an email from the iHeartChange website after the baseline questionnaires are complete.

At the 1 month and 6 month post enrollment, participants will receive the link to complete the questionnaire via email. Should they not complete the questionnaire within the first 2 weeks, they will receive reminder emails at 2, 4 and 6 weeks post initial send out. At the completion of the 1 month and 6 month questionnaires, the participant will receive a small incentive.

For all participants, a one-on-one telehealth session with the nurse will be set up. The session will take ~ 1 hour. Prior to the session the participant will receive a mail out transition package of additional written resources containing a "When You're 18 booklet" with transition specific information, disease specific information sheets, adolescent mental health resources, +/- endocarditis information if applicable.

Participant heart history information will be collected as well as demographics by accessing their paper charts, eClinician, Netcare and Connectcare electronic medical records. Baseline data we are collecting includes current height, weight, date of birth, cardiac diagnosis, cardiac surgery and procedure information, medications, cardiology visits and other information from the cardiology clinic letters.

DATA ANALYSIS:

Each participant will be assigned an alphanumerical code and pseudonym. All qualitative data (nursing logs, text/email transcripts) will be transcribed, anonymized, and analyzed for codes, categories and subcategories. The unit of analysis will be the nurse-led session; all data for each session will be analyzed together to get a sense of what happened, what influenced what happened, and whether the intervention was successful. Categories will be given descriptors that use words as close to the data as possible; eventually, categories will be grouped into main categories. Thematic analysis will be used to define broader categories of potential influences on intervention effectiveness with the unit of analysis being the entire set of coded session data.

The results of quantitative analyses will be compared with qualitative results to explore the extent to which there is agreement. Priority will be given to quantitative data; a nuanced understanding of what influenced intervention effectiveness will be sought through a process of integration.

ELIGIBILITY:
Inclusion Criteria:

* 16-25 year olds with moderate or complex congenital heart disease (CHD), as previously defined
* Followed in a cardiology satellite/outreach clinic affiliated with the Stollery Children's Hospital (High Level, Fort McMurray, Grand Prairie, Red Deer, Yellowknife)

Exclusion Criteria:

* less than a Grade 6 level of reading and comprehension, based on medical record review or parent report;
* heart transplantation, as this results in distinct health challenges.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
adolescents' knowledge of their heart | baseline, 1 month, 6 months
  Change in MyHeart Scale, between baseline, 1, and 6 months.

SECONDARY OUTCOMES:
Self-Efficacy | baseline, 1 month, 6 months
  Change in General Self-Efficacy (GSE) score between baseline, 1 and 6 months. GSE scores range from 0 to 40 with higher scores reflecting more self-efficacy.
Transition Readiness | baseline, 1 month, 6 months
  Change in Transition Q score between baseline, 1 and 6 months.
iHeartChange Use | 6 months
  The number of times participants have logged in to iHeartChange, and the number of pages within iHeartChange visited will be compared between the two study groups during the first 6 months post enrolment.
Nurse-adolescent Interactions | 6 months
  Qualitative data will consist of nurse-generated intervention logs and field notes recorded immediately following each session, and follow-up 7-day text messages/emails between study nurse and participants in the intervention group, detailing all nurse-adolescent interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mackie, MD, Principal Investigator — Stollery Children's Hospital
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No